CLINICAL TRIAL: NCT03681704
Title: Multicenter Clinical Study on the Treatment of Early Stage Diabetic Kidney Disease With Integrated Traditional Chinese and Western Medicine
Brief Title: the Integrated Traditional Chinese and Western Medicine Treat Early Stage DKD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17401970500-a
Record Dates: First submitted 2018-09-11; First posted 2018-09-24 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Diabetic Nephropathy Type 2
Keywords: Diabetic Kidney Disease，Traditional Chinese medicine
MeSH Terms: interventions — huangqi decoction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HuangQi Decoction (Experimental): HuangQi Decoction 150ml by mouth ,twice a day for 24 weeks
  Interventions: Drug: HuangQi Decoction
- HuangQi Decoction placebo (Placebo Comparator): HuangQi Decoction placebo 150ml by mouth, twice a day for 24 weeks
  Interventions: Drug: HuangQi Decoction placebo

INTERVENTIONS:
Drug: HuangQi Decoction — HuangQi Decoction 150ml twice a day for 24 weeks
  Other Names: Astragalus and other TCMs Decoction
  Arms: HuangQi Decoction
Drug: HuangQi Decoction placebo — traditional Chinese medicine placebo mimic HuangQi Decoction 150ml twice a day for 24 weeks
  Other Names: Astragalus Decoction placebo
  Arms: HuangQi Decoction placebo

SUMMARY:
Efficacy and Safety of treatment with Traditional Chinese Medicine HuangQi Decoctions in Patients with early stage of Diabetic Kidney Disease.

DETAILED DESCRIPTION:
The study is a multi-center, randomized, double-blind, placebo-controlled trial. It is performed in Longhua Hospital, Shanghai University of Traditional Chinese Medicine, Shanghai Jiao Tong University Affiliated Sixth People's Hospital, Putuo Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, and Shanghai Baoshan District Hospital of Integrated Traditional Chinese Medicine and Western Medicine, China.

ELIGIBILITY:
Inclusion Criteria:

1. Identify the diagnosis of type 2 diabetes;
2. It meets the medical history of diabetic kidney disease, according to the Mogensen diagnostic staging standard DKD III;
3. Age 18-75 years old, gender ＆ethnicity are not limited;
4. glycated hemoglobin ≤ 10%;
5. Blood pressure is controlled below 130/80mmHg

Exclusion Criteria:

1. Combine other ACEI and ARB application indications other than hypertension;
2. Combine severe primary diseases related to heart, brain, liver and hematopoietic system;
3. Patients who have acute metabolic disorders such as diabetic ketoacidosis occur in the past month;
4. Patients who HBV serological indicators except HbsAb are positive and persistent liver function test transaminase abnormalities;
5. Patients with malignant tumors or history of malignant tumors, history of HIV infection, history of psychosis, acute central nervous system diseases, severe gastrointestinal diseases, and banned use of immunosuppressive agents;
6. Patients with acute renal failure, combined with urinary tract infection, menstrual period, intense exercise, cold and other stress states;
7. pregnant or lactating women;
8. Patients who accepted other clinical trial studies on going ;
9. Patients who combined with serious diseases and dysfunctions in other organs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
ACR | 24 weeks
  the Urinary albumin/ creatinine ratios in stage Ⅲ diabetes kidney disease patients

CONTACTS AND LOCATIONS:
Overall Officials: Yueyi Deng, PhD, Principal Investigator — Shanghai University of Traditional Chinese Medicine
Locations (1):
- Longhua Hospital, Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality, China